CLINICAL TRIAL: NCT01844869
Title: An Open-Label Study to Investigate the Pharmacokinetics (Absorption, Distribution, Metabolism, and Excretion) of Omacetaxine Mepesuccinate Following Subcutaneous Administration of [14C]Omacetaxine Mepesuccinate in Patients With Relapsed and/or Refractory Hematologic Malignancies or Advanced Solid Tumors
Brief Title: An Open-Label Study to Investigate the Pharmacokinetics of Omacetaxine Mepesuccinate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C41443/1103 Study; 2012-004003-12 (EudraCT Number)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Hematologic Malignancies; Solid Tumors
Keywords: omacetaxine; omacetaxine mepesuccinate; pharmacokinetics; hematologic malignancies; advanced solid tumors
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- omacetaxine mepesuccinate (Experimental): Period A: 7-day pharmacokinetic assessment period in which all patients will be administered a single subcutaneous radiolabeled dose of 1.25-mg/m2 omacetaxine.
  Period B: omacetaxine will be administered as an sc injection at a dosage of 1.25 mg/m2 twice daily for 7 days (patients with solid tumors) or 14 days (patients with hematologic malignancies) of every 28-day cycle for up to 6 cycles.
  Interventions: Drug: omacetaxine mepesuccinate

INTERVENTIONS:
Drug: omacetaxine mepesuccinate
  Other Names: omacetaxine

SUMMARY:
The purpose of this study is to determine the pharmacokinetic and safety profiles of omacetaxine and its metabolites in patients with relapsed and/or refractory hematologic malignancies or advanced solid tumors following subcutaneous (sc) administration.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label, nonrandomized study to determine the pharmacokinetics (absorption, distribution, metabolism, and excretion) of omacetaxine and its metabolites following a sc dosage of 1.25 mg/m2 in adult patients with relapsed and/or refractory hematologic malignancies or advanced solid tumors. The study consists of a screening period of up to 28 days, followed by a 7-day pharmacokinetic assessment period (period A) that includes administration of a single radiolabeled dose of omacetaxine, an open-label treatment period of up to six 28-day cycles (period B), and a final assessment to occur approximately 28±7 days after the end of the last treatment cycle. Period B will begin after collection of the 72-hour pharmacokinetic sample during period A.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* The patient is at least 18 years of age at the time of informed consent.
* The patient has a histologically or cytologically confirmed diagnosis of any of the following:
* Relapsed or refractory leukemia, including Philadelphia chromosome-positive (Ph+), chronic myelogenous leukemia (CML), acute promyelocytic leukemia (APL), acute myelogenous leukemia (AML), or myelodysplastic syndrome (MDS).
* Advanced solid tumors (ie, breast, lung, head/neck, colorectal, melanoma, and sarcoma). The malignancy must be considered unresponsive to accepted available therapies.
* The patient has an estimated life expectancy of at least 3 months.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Other criteria apply.

Exclusion Criteria:

* The patient has had chemotherapy, radiotherapy, radioimmunotherapy, or immunotherapy within 28 days prior to the first dose of study drug or has not recovered from adverse events due to any agents administered previously. For patients who received therapy with mitomycin C, the interval is 42 days.
* The patient is receiving any other treatment for hematologic/nonhematologic malignancy.
* The patient has had previous treatment with omacetaxine.
* The patient has been treated with any hematopoietic growth factors within 14 days of study entry (patients on chronic erythropoiesis stimulating agents are allowed).
* The patient has New York Heart Association (NYHA) Class 3 or 4 heart disease, active ischemia, or any uncontrolled, unstable cardiac condition for which treatment for the condition is indicated but is not controlled despite adequate therapy, including angina pectoris, cardiac arrhythmia, hypertension, or congestive heart failure.
* The patient has experienced a myocardial infarction within the previous 12 weeks.
* The patient has a solid tumor with symptomatic central nervous system (CNS) metastases.
* The patient has an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
* Other criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentrations (Cmax) | 0,15, 30, and 45 minutes and 1, 2, 4, 8, 12, 24, 32, 48, 72, 96,120, 144, and 168 hours post dose
Time to Reach Maximum Observed Plasma Drug Concentration (Tmax) | 0,15, 30, and 45 minutes and 1, 2, 4, 8, 12, 24, 32, 48, 72, 96,120, 144, and 168 hours post dose
Area under the plasma concentration by time curve (AUC) from time 0 to infinity (AUC0-∞) | 0,15, 30, and 45 minutes and 1, 2, 4, 8, 12, 24, 32, 48, 72, 96,120, 144, and 168 hours post dose
Area under the Curve from Time Zero to the Time of the Last Measurable Drug Concentration (AUC0-t) | 0,15, 30, and 45 minutes and 1, 2, 4, 8, 12, 24, 32, 48, 72, 96,120, 144, and 168 hours post dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Terminal rate constant (λz) and associated half-life (t½) | 0,15, 30, and 45 minutes and 1, 2, 4, 8, 12, 24, 32, 48, 72, 96,120, 144, and 168 hours post dose
Percentage extrapolation calculated as (AUC0-∞-AUC0-t)/(AUC0-∞)x100 | 0,15, 30, and 45 minutes and 1, 2, 4, 8, 12, 24, 32, 48, 72, 96,120, 144, and 168 hours post dose
Apparent plasma clearance (CL/F) | 0,15, 30, and 45 minutes and 1, 2, 4, 8, 12, 24, 32, 48, 72, 96,120, 144, and 168 hours post dose
Apparent volume of distribution (Vz/F) | 0,15, 30, and 45 minutes and 1, 2, 4, 8, 12, 24, 32, 48, 72, 96,120, 144, and 168 hours post dose

SECONDARY OUTCOMES:
Summary of participants with adverse events | From Day 1 through the end of the follow-up period (28±7 days after 6 month treatment cycle)

CONTACTS AND LOCATIONS:
Locations (1):
- Teva Investigational Site 38045, Amsterdam, Netherlands